CLINICAL TRIAL: NCT06456645
Title: The Impacts of Maternal Smoking During Pregnancy on Breastfeeding and the Correlation of IGF, Leptin, HPL Expression in Placenta Tissue
Brief Title: Effects of Smoking on Placenta and Lactation
Status: Completed | Type: Observational
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Other Study IDs: MCBU_Smoking
Record Dates: First submitted 2024-05-29; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Smoking, Tobacco; Placenta Diseases; Breastfeeding; Fetal Conditions
Keywords: Smoking cigarette; placenta; IGF-1; Leptin; HPL; breastfeeding
MeSH Terms: conditions — Tobacco Smoking; Placenta Diseases; Breast Feeding; Cigarette Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Placenta tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1:: Smokers (study group)
- Group 2:: Non-Smokers (control group)

SUMMARY:
Maternal smoking during pregnancy although it is known to be associated with fetal growth restriction, it's effect on postpartum breastfeeding is not yet clear. The aim of the present study was to examine the impacts of smoking in pregnancy on breastfeeding as well as its impacts on placental immunoreactivity.

DETAILED DESCRIPTION:
The study was conducted on 70 women who gave birth via spontaneous vaginal delivery. Groups were classified as Smokers (n=35) and Non-smokers (n=35). The breastfeeding conditions of both groups were evaluated prior to discharge and after postpartum 10th day.

Cross-sections were taken from the placenta tissues after which their IGF-1 (insulin like growth factor-1), Leptin, HPL (human placental lactogen) immunoreactivities were examined.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who have started smoking at least 100 cigarettes in her lifetime and who now smokes every day,
* Pregnant women who have never smoked throughout their life, including pregnancy(16),
* Pregnant women who gave birth at term,
* Multiple pregnancy, preeclampsia, gestational diabetes, thyroid dysfunction, those who do not have a systemic disease and due to systemic disease during pregnancy those who do not use
* Pregnant women who had spontaneous vaginal delivery,
* In order not to encounter communication barriers and because cultural differences may vary, the pregnant woman is not a foreign national,
* Pregnant women who do not have any barriers to communication by phone,
* Those who do not have any health problems that prevent breastfeeding

Exclusion Criteria:

* multiple pregnancy
* insulin dependent diabetes
* pregnant women who have had a cesarean section
* preeclampsia
* thyroid disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant female
Study Population: Pregnant women who have started smoking at least 100 cigarettes in her lifetime and who now smokes every day
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
100% Patients's placenta with smoking in Pregnancy and 100% Patients's Placenta with from non-smoking in Pregnancy. Placenta Tissues Staining Measured by immunohistochemistry and biochemistry technique. | Baseline

SECONDARY OUTCOMES:
Sociodemographic, birth history, and breastfeeding questions were measured by survey technique. | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Manisa Celal Bayar Universitesi, Manisa, Turkey (Türkiye)